CLINICAL TRIAL: NCT02731547
Title: Education Against Tobacco: Medical-student-delivered Smoking Prevention Programme for Secondary Schools in Bosnia and Herzegovina - Randomized Trial
Brief Title: Education Against Tobacco Randomized Trial in Bosnia and Herzegovina
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Giessen (Other)
Collaborators: University of Dhaka (Other)
Responsible Party: Principal Investigator, Titus J. Brinker, cand. med. Titus J. Brinker, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCTBosnia
Record Dates: First submitted 2016-04-03; First posted 2016-04-07 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Tobacco Prevention; Tobacco; Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention group receives a school-based module taking about two hours delivered by medical students in the schools.
  Interventions: Behavioral: Education Against Tobacco School-Based Intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Education Against Tobacco School-Based Intervention
  Arms: Intervention group

SUMMARY:
A two armed randomized trial is evaluating the effect of the medical-student-delivered school-based intervention Education Against Tobacco on the smoking behavior of adolescents in 7-11th grade of secondary schools in Bosnia and Herzegovina. The primary endpoint is the change in smoking prevalence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Visiting grades 7-9 of regular secondary schools in Bosnia and Herzegovina.

Exclusion Criteria:

Not fulfilling inclusion criteria.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Smoking prevalence measured via questionnaire. | 12 months follow-up

SECONDARY OUTCOMES:
Smoking onset: Difference in the number of new smokers at 12 months of follow-up who were not present at baseline | Baseline and 12 months
Difference in the number of new non-smokers at 12 months of follow-up who were smoking at baseline | Baseline and 12 months
Relevant differences due to the theory of planned behaviour between the two groups measured via questionnaire. | Baseline and 12 months
  Difference in attitude towards smoking between the two groups at 12 months follow-up measured via questionnaires.

IPD SHARING:
Plan to Share IPD: Undecided